CLINICAL TRIAL: NCT01630187
Title: Comparison of Two Doses of Carbetocin for Prevention of Uterine Atony During Elective Cesarean Section: a Randomized Controlled Trial
Brief Title: Comparison of Two Doses of Carbetocin for Prevention of Uterine Atony, During Elective Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARB-011
Record Dates: First submitted 2012-05-17; First posted 2012-06-28 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Uterine Atony; Post-partum Hemorrhage
Keywords: Carbetocin; Uterotonic drug; elective cesarean section
MeSH Terms: conditions — Uterine Inertia; Postpartum Hemorrhage | interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbetocin 100 mcg (Active Comparator)
  Interventions: Drug: Carbetocin
- Carbetocin 50 mcg (Experimental)
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — Administration of carbetocin 50 mcg , after clamping the umbilical cord
  Arms: Carbetocin 50 mcg
Drug: Carbetocin — Administration of carbetocin 100 mcg , after clamping the umbilical cord
  Arms: Carbetocin 100 mcg

SUMMARY:
The purpose of this study is to evaluate the effectiveness of two doses of carbetocin (50 mcg vs 100 mcg) in preventing uterine atony during elective cesarean section.

DETAILED DESCRIPTION:
Postpartum hemorrhage is a major cause of mortality and morbidity in the world, and it is most often caused by uterine atony. To prevent this complication, uterotonic medication is used during elective cesarean section.

Carbetocin, a long-acting synthetic analogue of oxytocin, has been used for this purpose for many years. This medication has numerous side effects: hypotension, tachycardia, nausea, vomiting, chest pain, etc. Using a smaller dose of carbetocin might lower the incidence of these side effects, without compromising prevention of uterine atony in a low-risk group of patient.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* ≥ 37-week pregnancy
* singleton pregnancy
* elective cesarean section with a low transverse incision
* ASA I or II

Exclusion Criteria:

* Personal history of uterine atony or postpartum hemorrhage
* Abnormal placental implantation (known or suspected)
* > 3 cesarean sections in the past
* Personal history of a classic uterine incision
* Estimated fetal weight > 4500g
* Hemoglobin < 100 g/L
* Regular use of tocolytic drugs
* Cesarean section under general anesthesia
* Known allergy to carbetocin
* Refusal
* Inability to obtain informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Utilization of a second uterotonic drug | First 48 hours of the postpartum

SECONDARY OUTCOMES:
Incidence of side effects | During the fifteen minutes following the administration of carbetocin
Incidence of major complications | First 48 hours of the postpartum
Drop in hemoglobin measurement | on the second post-partum day

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bédard, Principal Investigator — Laval University
Locations (1):
- Hôpital Saint-François-d'Assise (CHUQ), Québec, Quebec, Canada